CLINICAL TRIAL: NCT06036719
Title: Interstitial Lung Disease: A Study From Infancy to Elderly Including Relatives
Acronym: RaDiCo-ILD 2
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-58; 2021-A00094-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-08-03; First posted 2023-09-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Interstitial Lung Diseases
Keywords: Pediatric Interstitial Lung Diseases; Idiopathic Pulmonary Fibrosis; Pediatrics / adult; Idiopathic Interstitial Pneumonia
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Idiopathic Interstitial Pneumonias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The concerned patients are children and adults suffering from idiopathic interstitial pneumonias, other chronic fibrosing interstitial pneumonias with a progressive phenotype, and interstitial pneumonia associated with Scleroderma and related cases of patients carrying a mutation on one of the telomere-associated genes.

This is a national, observational, longitudinal, multicenter study that will be conducted retrospectively and prospectively. It aims to collect consistent and comparable clinical data for patients and their relatives, whether they carry a mutation or not, affected by diffuse idiopathic interstitial pneumopathy.

The expected duration of the study, including data analysis, is approximately 10 years (5 years for participant enrollment and 5 years of follow-up, in addition to the steps for data management and statistical analyses).

Each participating center will inform every participant by providing an information sheet, and their written consent will be obtained before including them in the study and commencing data collection.

Prospective medical data will be collected at 6 months to 1 year after enrollment and then at least once per year for patients up to 5 years and 5 years for their relatives.

Participants will complete a self-questionnaire during their regular follow-up consultations or by accessing a secure interface.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of IIP established based on clinical, radiological, or functional criteria.

Confirmed diagnosis of non-IPF progressive fibrotic interstitial lung disease (PF-ILD) with fibrosis ≥ 10% on CT scan, disease worsening not related to pulmonary embolism, decompensated heart failure, or lower respiratory tract infection, and disease progression despite "appropriate management" evaluated over a period of up to 24 months:

* A relative decline in Forced Vital Capacity (FVC) of at least 10% from predicted value, with or without clinical deterioration, or
* A combination of at least 2 of the following criteria: a relative decline in FVC between 5% and 10% from predicted value, worsening respiratory symptoms, increased extent of pulmonary fibrosis on thoracic CT scan.

Confirmed diagnosis of Systemic Sclerosis-associated Interstitial Lung Disease (SSc-ILD) (American College of Rheumatology criteria), with a total score ≥ 9 and disease extent involving ≥ 10% of the lungs (defined by reticular abnormalities, honeycombing, and ground-glass opacities) on high-resolution CT (HRCT) scan.

For relatives: First degree relatives of patients carrying a mutation in TERT, TERC, RTEL1, TINF2, DKC1, PARN genes, and other telomere related genes that may be described in the future and included.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study cohort will include:
  * Prevalent and incident cases of symptomatic adult and paediatric patients with a diagnosed IIP, other chronic fibrosing ILDs with progressive phenotype, SSc-associated ILDs. In total, 2850 patients are expected. 1600 patients are already included via the initial protocol RaDiCo-PID.
  * Cases corresponding to patients included as 1st degree relatives of a symptomatic diagnosed FPF patient carrying a specific mutation. About 150 relatives are expected in this protocol. No inclusion in initial protocol because it is a new population.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2031-03-19 (Estimated); Study Completion 2031-03-19 (Estimated)

PRIMARY OUTCOMES:
Family history | At inclusion visit
Clinical parameters : respiratory examination | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Collection of biological parameters | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Chest scan | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Chest radiographs | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Pulmonary scintigraphy | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Chest RMI | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Echocardiography | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Search for infectious agents | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Bronchoscopy | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Lung function tests: Arterial blood gas | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Lung function tests: if available sleep gas exchange | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Lung function tests: polysomnography | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Lung tissue examination, if available Lung biopsy (surgical, transbronchial), Lung explant, if lung transplant | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Assessment of digestive function | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Assessment of cardiac function (cardiovascular ultrasound) | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Assessment of cardiac function (cardiac magnetic resonance imaging) | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Assessment of cardiac function ( right heart catheterization) | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Dermatological evaluation | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Fertility evaluation | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Bone densitometry | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Collection of patient treatments | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients
  treatment name, dosage, start and end dates..

SECONDARY OUTCOMES:
Genetic assessment | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
  Identification of gene factors involved in disease initiation and progression
The description of data on environmental and co-morbidity factors impacting disease severity | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Validate already published biomarkers candidates for disease diagnosis | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Validate already published biomarkers candidates for disease progression. | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
SARS-CoV2: Method of diagnosis, symptoms, medical supports, treatments | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Immuno-hematological assessment | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
  Presence of macrocytosis, thrombocytopenia, anaemia, dysmyelopoiesis, myelodysplasia, aplasia, or acute leukaemia
Hepatic assessment (hepatocellular carcinoma) | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
  Liver function tests, cirrhosis, hepatocellular carcinoma
Hepatic assessment (Liver function tests) | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Hepatic assessment (cirrhosis) | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Cutaneous assessment | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Pulmonary emphysema on the thoracic scanner and evaluated by double reading of the scanner | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Spermogram assessment | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Hormonal evaluation | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Osteopenia, osteoporosis | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives
Solid cancer including skin cancer and cervical dysplasia (current cancer and history of cancer) | Through study completion, at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year for patients, and at inclusion and 5 years for relatives

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Cottin, Pr, Principal Investigator — Centre National de Référence des maladies pulmonaires rares
Locations (1):
- RaDiCo-ILD2, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided